CLINICAL TRIAL: NCT04167488
Title: Assessment of Physical Activity Among Juvenile Idiopathic Arthritis Children Performed With Actigraphy
Acronym: AJIACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2019/432
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Actigraphic measurement (Experimental)
  Interventions: Device: Actigraphic measurement

INTERVENTIONS:
Device: Actigraphic measurement — Physical activity assessed with actigraphic device worn during 7 days

SUMMARY:
This study aims to describe physical activity among juvenile idiopathic arthritis children, according to the disease's and patient's characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile idiopathic arthritis evolving for more than a year

Exclusion Criteria:

* intra-articular infiltration performed less than a month ago

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity assessment | Day 7
  Physical activity will be measured with actigraphic device and children will be divided into 3 groups of activity levels: low / moderate / high.
  Low is < or = 1000 counts per minute Moderate is > 1000 counts per minute High is > 2500 per minute

CONTACTS AND LOCATIONS:
Overall Officials: Claire BALLOT SCHMIT, MD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No